CLINICAL TRIAL: NCT06485804
Title: Comparing Efficacy and Adherence of Smartphone-guided Exercises to Conventional Self-directed Exercises for Neck Pain in Office Workers: A Randomized Controlled Trial Protocol
Brief Title: AI Mobile App vs Self Exercises in Workers With Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Collaborators: Sana Salah (Unknown); Amr Chaabeni (Unknown)
Responsible Party: Principal Investigator, Anis Jellad, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIMobApp-Neck-Pain
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Work-Related Condition
Keywords: Office Workers; Clinical trial Protocol; Exercise Therapy; Mobile Application; Neck Pain; Patient compliance; Self-management; Workplace
MeSH Terms: conditions — Neck Pain; Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will use a smartphone application which will provide an individualized exercises program.
  Interventions: Other: Smartphone application guided exercises
- Control group (No Intervention): Participants in the control group will receive a rehabilitation program delivered on a paper sheet containing pictures of exercises with written explanations in French, including the number of sets and repetitions

INTERVENTIONS:
Other: Smartphone application guided exercises — Participants in the intervention group will use a smartphone application to execute a self-rehabilitation program. The app will integrate:
  * Basic information about neck pain and ergonomic advice.
  * A series of evaluation questions on pain and function.
  * Appropriate sets of exercises with videos and instructions.
  * Daily reminders.
  * Evaluation reports providing feedback and adherence.
  Arms: Intervention group

SUMMARY:
This study aims to compare the impact of two different methods to administer self-exercises in administrative workers with neck pain: an Artificial Intelligence embedded mobile application and written sheet.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a chronic NP lasting for more than three months, and a pain level at baseline assessment ≥ 30 (VAS)

Exclusion Criteria:

* Acute neck pain, neck pain from specific causes (eg; Chronic inflammatory diseases), spine trauma or surgery, cervical radiculopathy or myelopathy, and physical therapy treatments in the last six months before baseline assessment.

Ages: 30 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Pain intensity will be assessed at baseline, and at 4, and 8 weeks of follow-up.
  Pain intensity assessed using a Visual Analog Scale on a scale from 0 to 100.

SECONDARY OUTCOMES:
Function | Function will be assessed at baseline, and at 4, and 8 weeks of follow-up.
  Patient function will be assessed using the neck disability index (NDI). The scale consists of a set of questions addressing various aspects of neck pain and its influence on activities such as personal care, lifting, reading, working, and recreation
Quality of life measure | Quality of life will be assessed at baseline, and at 4, and 8 weeks of follow-up.
  The short form 12 (SF-12) will be used to measure health-related Quality of life. The SF-12 is a shorter version of the short form 36 (SF-36) and is used to assess individual's physical and mental well-being.
Patient adherence | Patient adherence will be assessed at 4, and 8 weeks of follow-up.
  Adherence will be measured using a frequency-based response scale (ie; never, seldom, often, almost always, and always) adapted from the adherence scale of Sluijs et al. (Phys Ther 1993)

OTHER OUTCOMES:
Gender | Assessed at baseline
  Gender: Female, Male.
Age | Assessed at baseline
  Age in terms of years
Body mass index (BMI) | Assessed at baseline
  BMI is calculated as follows: BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height (in metres) squared.
Comorbidities | Assessed at baseline
  Comorbidities comprise: Diabetes, Hypertension, Thyroid disorders, Cardiovascular and Lung diseases, and Cancer history.
Musculoskeletal disorders | Assessed at baseline
  Musculoskeletal disorders comprise: Osteoarthrities, Rheumatic arthritis, Osteoporosis, and Tendinopathies.
Work seniority | Assessed at baseline
  Work seniority: Length of work service (years).
Time spent in front of computer | Assessed at baseline
  Time spent in front of computer: average number of daily hours spent in front of computer.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Salah, Professor, Principal Investigator — University of Monastir

REFERENCES:
- [Derived] Salah S, Jellad A, Mili M, Chaabeni A, Bedoui MH, Ben Saad H. Comparing efficacy and adherence of smartphone-guided exercises to conventional self-directed exercises for neck pain in office workers: A randomized controlled trial protocol. PLoS One. 2025 Sep 19;20(9):e0329863. doi: 10.1371/journal.pone.0329863. eCollection 2025. PMID 40971708